CLINICAL TRIAL: NCT00250575
Title: A 24-week, Multicenter, Open-label Study to Evaluate the Safety and Efficacy of Clozapine in Patients With Treatment-resistant Schizophrenia
Brief Title: A Study to Evaluate the Safety and Efficacy of Clozapine in Patients With Treatment-resistant Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLEX123J1301
Record Dates: First submitted 2005-11-07; First posted 2005-11-08 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia, treatment-resistant, clozapine
MeSH Terms: conditions — Schizophrenia | interventions — Clozapine

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Clozapine

INTERVENTIONS:
Drug: Clozapine
  Other Names: Clozaril

SUMMARY:
Clozapine is an antipsychotic. This 24-week study will evaluate the safety and efficacy of clozapine in patients with treatment-resistant schizophrenia.

This study is not recruiting in the United States.

DETAILED DESCRIPTION:
Clozapine is an antipsychotic. This 24-week study will evaluate the safety and efficacy of clozapine in patients with treatment-resistant schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as schizophrenia
* Not responded to at least two atypical antipshychotics launched in Japan
* Inpatient

Exclusion Criteria:

* Low white blood cell count
* Significant heart diseases
* Diabetes mellitus

Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2005-11; Primary Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Values of hematological tests during the 24 week treatment
Incidence of hematological adverse events during the 24 week treatment
Compliance to Clozapine Patient Monitoring System during the 24 week treatment

SECONDARY OUTCOMES:
Changes in the symptoms of psychosis every 4 weeks up to week 24
Global change in severity of psychosis at baseline and week 12
Global impression of change in the condition of patients at week 12 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (8):
- Japan (8):
  - Novartis Investigational Site, Chiba
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Ishikawa
  - Novartis Investigative Site, Osaka
  - Novartis Investigative Site, Saga
  - Novartis Investigative Site, Tokyo
  - Novartis Investigative Site, Toyama
  - Novartis Investigative Site, Yamanashi